CLINICAL TRIAL: NCT02619591
Title: Comparison Of Chest Ultrasound Techniques To Identify Clinically Significant Pneumothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Executive Vice Chairman, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Umass
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2015-12

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Imaging - Single View (Active Comparator): Ultrasound performed on patient. A single view of each hemithorax with ultrasound was performed on patient
  Interventions: Other: Ultrasound Imaging
- Ultrasound Imaging - Multiple Views (Experimental): Ultrasound performed on patient. Multiple view of each hemithorax with ultrasound was performed on patient
  Interventions: Other: Ultrasound Imaging

INTERVENTIONS:
Other: Ultrasound Imaging — views of a hemithorax was obtained using the Zonare Ultrasound machine.

SUMMARY:
Patients with chest trauma undergo ultrasound to detect a collapsed lung. Two techniques have been described. A single view for each hemi-thorax, and multiple views for each hemithorax. The investigators are comparing these two techniques in a randomized prospective trial.

DETAILED DESCRIPTION:
This is a randomized, prospective blinded study on trauma patients arriving to an emergency department.

Study Setting and Population This study will be conducted on the University Campus of the University of Massachusetts Medical Center, which is an urban academic emergency department that sees 80,000 patients annually and has a dedicated Level I trauma service that is staffed by trauma surgery and emergency medicine. Adult patients with acute traumatic injury who are undergoing a CT scan of the chest are eligible for enrollment.

Study Protocol Trauma patients are enrolled as they arrived to the emergency department. The investigators will include any trauma patient aged 18 and over. The investigtors will exclude any patient who was too unstable and required clinical care that prevented performing a chest wall ultrasound, patients with a chest tube in place prior to arrival, pregnant women, and prisoners. Imaging decisions on trauma patients will be made early on in their evaluation. The patient will be assigned using a pre-determined randomization scheme to a single view or four views of each hemi-thorax prior to any imaging being done. Ultrasounds will be performed and interpreted by credentialed physicians using a 7.5Mhz linear array transducer on a portable ultrasound machine (Zonare z.one ultra) with digital clips recorded for later review. When the investigators obtain a single view of each hemi-thorax, the probe will be placed in a longitudinal orientation on the midclavicular line in the third intercostal space. When the investigators obtain four views of each hemi-thorax, the first image location will be the same as in the single view and then the probe will be moved inferiorly and laterally to obtain the additional three images. Immediately following the ultrasound examination, the patient will be transported to the CT scanner for further imaging.

The goal of this study is to determine if a single view of each hemi-thorax can identify a pneumothorax or if additional images should be included. The primary study endpoint is the presence of a pneumothorax on ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had trauma and are receiving a chest CT.

Exclusion Criteria:

* Clinically Unstable
* Clinical care prevented ultrasound
* Patient with a chest tube in place
* Pregnant Women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, Principal Investigator — UMASS Memorial

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with chest trauma presenting to the emergency department who were going to get a CT of the chest were eligible
Pre-assignment Details: Exclusions were patients who had recieved a chest tube already, or those with known pneumothoraces.
Groups:
- "Device" - Ultrasound Imaging - Single View: Ultrasound performed on patient. A single view of each hemithorax with ultrasound was performed on patient
  Ultrasound Imaging Technique - Single View: A single view of a hemithorax was obtained using the Zonare Ultrasound machine.
- "Device" - Ultrasound Imaging - Multiple Views: Ultrasound performed on patient. Multiple view of each hemithorax with ultrasound was performed on patient
  Ultrasound Imaging Technique - Multiple Views: Multiple views of a hemithorax was obtained using the Zonare Ultrasound machine.
Period: Overall Study
Arm/Group | "Device" - Ultrasound Imaging - Single View | "Device" - Ultrasound Imaging - Multiple Views
Started | 139 | 121
Completed | 0 | 0
Not Completed | 139 | 121

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Imaging - Single View | Ultrasound Imaging - Multiple Views | Total
Number analyzed (Participants) | 139 | 121 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13) | 45 (12) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 100 | 86 | 186
Region of Enrollment [Number; unit: participants]
  United States | 139 | 121 | 260
Blunt Trauma [Number; unit: participants]
  Blunt Truama | 133 | 115 | 248
  Penetrating Trauma | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pneumothorax (Positive or Negative)
Description: The presence of a pneumothorax at the time of the ultrasound
Time Frame: up to 20 minutes
Measure: Number; unit: participants
Arm/Group | "Device" - Ultrasound Imaging - Single View | "Device" - Ultrasound Imaging - Multiple Views
Number analyzed (Participants) | 139 | 121
participants | 17 | 21

ADVERSE EVENTS:
Time Frame: 1 week
Description: Truama patients were followed for their admission time
Arm/Group | "Device" - Ultrasound Imaging - Single View | "Device" - Ultrasound Imaging - Multiple Views
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/121
Other Adverse Events (participants affected / at risk) | 0/139 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes